CLINICAL TRIAL: NCT04226391
Title: Surgical Flow Disruptions Inside the Operating Room, Intra-operative Teamwork, Stress and Post-operative Patient-outcomes: An Observational Study
Brief Title: Interruptions, Teamwork, Stress and Patient Outcomes in the Operating Room
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Matthias Weigl, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: FD&OUTCOME01
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Intraoperative Flow Disruptions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RAS Partial Nephrectomy
- RAS Radical Prostatectomy

SUMMARY:
The operating theatre (OR) in hospitals is a highly complex working environment and can withstand a variety of stresses and strains for the surgical team. So-called "Flow Disruption Events" (FDs) with a potential risk to patient safety occur very often.

The aim of the planned study project is to determine the effects of flow disruption events in the operating theatre on patients, the OR team and the duration of the surgery. The investigators plan an observational study at two university hospital in Southern Germany. The study population includes the entire surgical team during selected surgical procedures as well as the patients treated. The planned sample size is 82 surgical procedures. The investigators intend to collect data in two surgical specialties: Urology and traumatology.

Selected surgeries are evaluated by a trained observer and the interruptions and distractions in the course of the surgery are observed with a standardized tool. In addition, non-technical skills of the OR team are recorded: all members of the OR team will complete a short standardized questionnaire that measures mental workload and stress during the procedure. Additionally, post-operative patient outcomes are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Written consent, completed case
* OR Team: Written consent, at least 3 months working experience in the clinic, present for the majority of the procedure duration

Exclusion Criteria:

- OR visitors & students

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery in one of the participating departments
  Surgical teams including surgeons, nurses and anesthetists
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative Teamwork | 4 Hours
  Teamwork within the medical team including surgeons, nurses and anaesthetists
Stress, Mental Workload | 4 Hours
  Intraoperative workload, perceived distraction and stress of medical team
Patient Outcomes | 3 Months
  Intra- and postoperative patient outcomes (Complications, functional outcomes etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Urological Clinic and Outpatient Clinic, University hospital of the Ludwig-Maximilians-University (LMU) Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch A, Quartucci C, Buchner A, Schlenker B, Becker A, Catchpole K, Weigl M. Associations of flow disruptions with patient, staff, and process outcomes: a prospective observational study of robotic-assisted radical prostatectomies. Surg Endosc. 2023 Sep;37(9):6964-6974. doi: 10.1007/s00464-023-10162-2. Epub 2023 Jun 19. PMID 37336845